CLINICAL TRIAL: NCT07189559
Title: Digital Bodies: A Brief Intervention in Secondary Schools to Reduce Negative Body Image Among Adolescents in the Digital Age
Brief Title: School-Based Body Image Concerns Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Villa Garda Hospital (Other)
Responsible Party: Principal Investigator, Riccardo Dalle Grave, Head nutrition and endocrinology Villa Garda Hospital, Villa Garda Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: D.BODY/2025
Record Dates: First submitted 2025-09-16; First posted 2025-09-24 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Wait List Control; Intervention Program
Keywords: school-based intervention; adolescents; unrealistic appearance ideals; social media

STUDY DESIGN:
Intervention Model Description: Intervention vs no intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital Bodies intervention (Experimental): The Digital Bodies intervention consists of a one-hour interactive session. The session begins with a brief self-affirmation exercise, in which participants are asked to describe something important to them and explain why.
  The core of the intervention involves the use of cognitive dissonance techniques and the development of critical literacy skills to encourage adolescents to critically reflect on appearance ideals, as well as to foster the skills needed to challenge such ideals.
  The content focuses on (i) the socially constructed nature of body ideals across time and culture, with particular attention to social media spaces, (ii) the deconstruction of myths surrounding the "perfect body" (e.g., image editing, idealization), again with a focus on social media environments, and (iii) the role of adolescents in creating, perpetuating, and reinforcing these ideals through digital technologies, including social media.
  Interventions: Behavioral: Digital Bodies
- Waitlist control (No Intervention): No-intervention control group. To ensure that all students benefit from the intervention, the control group received the intervention after the 8 weeks.

INTERVENTIONS:
Behavioral: Digital Bodies — The Digital Bodies intervention consists of a one-hour interactive session. The core of the intervention involves the use of cognitive dissonance techniques and the development of critical literacy skills to encourage adolescents to critically reflect on appearance ideals, as well as to foster the skills needed to challenge such ideals.
  Arms: Digital Bodies intervention

SUMMARY:
The present study, sought to adapt Digital Bodies (a single-session intervention promoted in the United Kingdom (Bell et al., 2022) for the Italian school context and to assess its effectiveness as a single-session intervention aimed at challenging unrealistic appearance ideals and appearance-related pressures within social media environments. The study includes a cluster randomized controlled trial with two assessment points (baseline, post-intervention and 8-week follow-up) comparing the "Digital Bodies" program to a no-intervention control group. To ensure that all students benefit from the intervention, the control group received the intervention after the 8 weeks.

DETAILED DESCRIPTION:
The investigators conducted a cluster randomized controlled trial with two assessment points (baseline, post-intervention and 8-week follow-up) comparing the "Digital Bodies" program to a no-intervention control group. To ensure that all students benefit from the intervention, the control group received the intervention after the 8 weeks.

Randomization was performed at the school level, not the student level. This is known as cluster randomization, and it aims to avoid "contamination effects" (Smolak & Levine, 2001).

The research protocol was approved by the GHC Institutional Review Board (Protocol No. 0025GHCIRB). Written informed consent was obtained from each participant and their parent(s) or legal guardian(s), authorizing the collection and anonymized use of data for research purposes.

Participants Four hundred and forty-nine eligible participants were recruited from December 2024 to May 2025. Secondary school administrators were approached either by phone or email and received an information letter describing the key elements of the prevention program. Participation required the school principal-or a designated representative-to provide written confirmation through a signed agreement. Eligible participants were students in their first or second year of upper secondary school who, along with their parents, provided written informed consent. Students who did not complete the baseline questionnaire and the case report form were excluded from the analysis but were still permitted to participate in the intervention itself.

The "Digital Bodies" Program and Study Implementation The Digital Bodies intervention, adapted from an English study that demonstrated its effectiveness (Bell et al., 2022), consists of a one-hour interactive session. The session begins with a brief self-affirmation exercise, in which participants are asked to describe something important to them and explain why. When used at the start of the intervention, this technique can help reduce participants' initial resistance to health-promotion messages.

The core of the intervention involves the use of cognitive dissonance techniques and the development of critical literacy skills to encourage adolescents to critically reflect on appearance ideals, as well as to foster the skills needed to challenge such ideals.

The content focuses on (i) the socially constructed nature of body ideals across time and culture, with particular attention to social media spaces, (ii) the deconstruction of myths surrounding the "perfect body" (e.g., image editing, idealization), again with a focus on social media environments, and (iii) the role of adolescents in creating, perpetuating, and reinforcing these ideals through digital technologies, including social media.

The session concludes with an implementation-intentions exercise, where participants develop specific behavioral plans describing how they would act in three situations in which appearance ideals are most salient, to challenge or resist them.

ELIGIBILITY:
Inclusion Criteria:

* First or second year of upper secondary school

Exclusion Criteria:

* They and their parents did not provide written informed consent

Ages: 13 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 449 (Actual)
Dates: Start 2024-11-06 (Actual); Primary Completion 2025-05-29 (Actual); Study Completion 2025-05-29 (Actual)

PRIMARY OUTCOMES:
Body Satisfaction | Basal, post.treatment, 8-week follow-up
  Body satisfaction was measured using the Body Satisfaction Scale (BSS) (Bird et al., 2013). The scale comprises five items (e.g., "Do you feel satisfied with your appearance?"), rated on a 5-point Likert scale (1 = never, 5 = very often). Total scores range from 1 to 25, with higher values indicating greater body satisfaction. The items were translated into Italian and back-translated by a professional bilingual.
Internalization of Appearance Ideals | Basal, post-intervention, 8-week follow-up
  Internalization of appearance ideals was assessed using the Sociocultural Attitudes Towards Appearance Questionnaire (SATAQ-4R). The SATAQ-4R, in both its male and female forms, consists of seven conceptually coherent subscales. Three of these capture aspects of internalization. The remaining four subscales assess perceived sociocultural pressures: from family, peers, significant others, and the media.
  Each item is rated on a 5-point Likert scale (1 = strongly disagree, 5 = strongly agree). Higher scores indicate higher perceived sociocultural pressures
Self-Objectification | Basal, post-intervention, 8-week follow-up
  Self-objectification was evaluated with the Likert Self-Objectification Questionnaire (LSOQ) (Wollast et al., 2021). Participants ranked 10 body attributes according to their importance for self-concept (1 = not at all important, 11 = very important). Five attributes reflect appearance (e.g., sexual appeal, physical attractiveness), while five reflect competence (e.g., health, strength). Scores are calculated by subtracting the sum of the appearance attributes from the sum of the competence attributes (range= -25 to 25). Higher scores reflect a greater emphasis on the importance of appearance-based physical attributes over competency-based attributes, that is, high levels of self-objectification.

CONTACTS AND LOCATIONS:
Locations (1):
- Villa Garda Hospital, Garda, Verona, Italy

IPD SHARING:
Plan to Share IPD: No